CLINICAL TRIAL: NCT06842940
Title: Evaluating Slew Rate As a Predictor for Optimal Lead Fixation in Transvenous Cardiac Implantable Devices: a Prospective Multicenter Study
Brief Title: Slew Rate As a Predictor for Optimal Lead Fixation
Acronym: SLEW REGISTRY
Status: Recruiting | Type: Observational
Sponsor: Paolo Pastori, MD (Other)
Collaborators: University Hospital of Ferrara (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Sponsor-Investigator, Paolo Pastori, MD, Paolo Pastori, MD, Azienda Unità Sanitaria Locale di Parma
Organization: Azienda Unità Sanitaria Locale di Parma (Other)
Other Study IDs: 920/2021/OSS/AUSLPR
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Defibrillators, Implantable; Electrodes, Implanted; Pacemaker, Artificial; Predictive Value of Tests
Keywords: pacemaker; implantable cardiac defibrillator; lead; slew rate; sensing; active fixation; electrical performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients: Patients undergoing a transvenous cardiac devices implant with active lead fixation (pacing or defibrillator leads)

SUMMARY:
The goal of this observational study is to identify the most reliable electrical parameter measured at the time of implantation that can predict optimal lead fixation and long-term lead performance in patients undergoing transvenous pacemaker or implantable cardioverter-defibrillator (ICD) implant.

The main questions it aims to answer are:

* Is there a correlation between the slew rate measured at the time of lead implantation and the sensing measured at the 12-month follow-up?
* Is there a correlation between all electrical parameters recorded at implantation (including slew rate, current of injury, acute sensing, acute impedance, and acute pacing threshold) and the electrical parameters assessed at 12 months post-implantation (specifically chronic sensing, chronic impedance, and chronic pacing threshold)? Participants will undergo regular follow-up evaluations, with device interrogation visits scheduled at 1 and 12 months post-implantation as part of routine clinical care.

DETAILED DESCRIPTION:
During the implantation of transvenous pacemakers and implantable cardiac defibrillators, the placement of active fixation leads requires the measurement of standard electrical parameters (sensing, impedance, and capture threshold) to identify the optimal pacing site before helix deployment into the cardiac muscle. Selecting the optimal site at the time of implantation is crucial to ensure long-term lead performance and to prevente potential device malfunctions secondary to threshold elevation or sensing reduction.

Two additional electrical parameters-slew rate and the current of injury-may aid in selecting the optimal pacing site. However, these parameters have been poorly studied in the literature and exhibit significant differences. While the slew rate is easily measurable, as it is automatically determined by the pacing system analyzer (PSA), the current of injury requires non-standardized, complex, operator-dependent, and time-consuming manual measurements. Additionally, the slew rate can be assessed before helix deployment, whereas the current of injury can only be measured after helix fixation. While the current of injury generally indicates adequate helix fixation, at least in the acute setting, the significance of slew rate in predicting long-term lead stability remains uncertain.

The study hypothesis is that the slew rate significantly correlates with sensed electrical activity at 12 months post-implantation and may therefore serve as a predictor of optimal long-term lead fixation and performance.

This is a prospective, observational, single-arm, investigator-initiated, multicenter, non-profit cohort study. Four Italian centers are participating: Ospedale di Fidenza, Arcispedale Santa Maria Nuova di Reggio Emilia, Ospedale Civile di Piacenza, and Azienda Ospedaliero-Universitaria di Ferrara.

Patients undergoing pacemaker or ICD implantation with active-fixation atrial or ventricular leads, either for pacing or defibrillation, will be enrolled. The lead fixation site (right ventricular apex or septum) and pacing modality (traditional right ventricular pacing or conduction system pacing) will be determined at the physician's discretion.

Electrical parameters at implantation-including slew rate, current of injury, sensing, impedance, and capture threshold-will be measured in all participating centers using the same pacing system analyzer (PSA) model (Medtronic, Model 2290). Slew rate, sensing, impedance, and capture threshold will be assessed before and after helix deployment, as well as after lead fixation.

The current of injury is defined as an increase in ST-segment elevation of at least 5 mV for ventricular leads and 1 mV for atrial leads compared to baseline in the intracardiac electrogram (EGM).

All characteristics of the current of injury-including total intracardiac EGM duration, maximum ST elevation, and maximum ST elevation 80 msec after the first EGM deflection-will be assessed immediately after helix deployment, as the current of injury is a dynamic and time-dependent electrical phenomenon.

Following implantation-after device connection and prior to discharge-and throughout the follow-up period, electrical parameters (sensing, impedance, and capture threshold) will be assessed using the device programmer provided by the manufacturer of the implanted device.

Follow-up visits are scheduled at 1 and 12 months post-implantation and may be conducted either as in-person ambulatory visits or via remote monitoring, according to the standard clinical practice of each center. During these visits, lead dislodgement and any significant variations in electrical parameters will also be assessed. The total follow-up duration is 12 months from implantation.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of a transvenous pacemaker with active lead fixation.
* Implantation of a transvenous implantable cardioverter-defibrillator (ICD) with active lead fixation.

Exclusion Criteria:

* Pregnancy.
* Age under 18 years.
* Implantation of a subcutaneous ICD (S-ICD).
* Implantation of a leadless pacemaker.
* Patients requiring a new lead position with a previously implanted pacemaker or ICD

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with an indication for scheduled or urgent transvenous pacemaker or implantable cardioverter-defibrillator (ICD) implantation with active lead fixation
Sampling Method: Non-Probability Sample
Enrollment: 516 (Estimated)
Dates: Start 2023-02-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Slew rate value of active fixation leads (pacing or defibrillator leads) measured at the time of implantation | After the enrollment, at the time of implantation, prior to helix deployment for active lead fixation
  The slew rate value of active fixation leads (pacing or defibrillator leads) measured at the time of implantation will be automatically measured in millivolts (mV) using a Medtronic pacing system analyzer (PSA) (Model 2290) prior to helix deployment for active lead fixation. Both pacemaker and implantable cardioverter-defibrillator (ICD) leads will be included in the study. The lead fixation site (right ventricular apex or septum) and the implantation approach (traditional pacing or conduction system pacing) will be determined at the physician's discretion.

SECONDARY OUTCOMES:
Current of injury of active fixation leads (pacing or defibrillator leads) measured at the time of implantation | After the enrollment, at the time of implantation, immediately following helix deployment for active lead fixation
  Characteristics of the current of injury-including total intracardiac EGM duration (msec), maximum ST elevation (mm), and maximum ST elevation 80 msec after the first EGM deflection (mm)-will be manually measured using the Medtronic PSA Model 2290 immediately after helix deployment during implantation
Sensing of active fixation leads (pacing or defibrillator leads) | From enrollment at the time of implantation to the end of follow-up at 12 months
  Sensing (mV) will be automatically measured using the PSA 2290 before and after helix deployment, as well as after lead fixation, followed by assessment via the device programmer at the end of the implant procedure and prior to discharge.
  During scheduled device interrogation visits at 1 and 12 months post-implant, sensing will be evaluated automatically using the device programmer.
Capture threshold of active fixation leads (pacing or defibrillator leads) | From enrollment at the time of implantation to the end of follow-up at 12 months
  Capture threshold (volts with a fixed impulse duration of 0.4 msec) will be manually measured using the PSA 2290 before and after helix deployment, as well as after lead fixation. This will be followed by assessment via the device programmer at the end of the implant procedure and prior to discharge.
  During scheduled device interrogation visits at 1 and 12 months post-implant, capture threshold will be manually evaluated using the device programmer.
Impedance of active fixation leads (pacing or defibrillator leads) | From enrollment at the time of implantation to the end of follow-up at 12 months
  Impedance (ohm) will be automatically measured using the PSA 2290 before and after helix deployment, as well as after lead fixation, followed by assessment via the device programmer at the end of the implant procedure and prior to discharge.
  During scheduled device interrogation visits at 1 and 12 months post-implant, impedance will be evaluated automatically using the device programmer.

OTHER OUTCOMES:
Lead dislodgement | From the implantation to the end of follow-up at 12 months
  Any lead dislodgement (0 = No; 1 = Yes) occurring within the first 12 months post-implantation will be documented
Significant variation in electrical parameters | From the implantation to the end of follow-up at 12 months
  Any significant variation in electrical parameters occurring within the first 12 months post-implantation during follow-up will be documented, defined as follows:
  Pacing threshold: increase of >1.5 V (with a fixed impulse duration of 0.4 msec) Sensing: decrease to <4 mV Impedance: increase to >1500 ohms

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pastori, MD, Principal Investigator — Cardiology Unit, Medical and Diagnostics Department, Fidenza Hospital, Azienda USL of Parma
Locations (1):
- Azienda Unità Sanitaria Locale di Parma, Fidenza, Italy

IPD SHARING:
Plan to Share IPD: No